CLINICAL TRIAL: NCT01239043
Title: Antibody Persistence and Response to Re-vaccination With Either Menactra® or Menomune® Vaccine Approximately Three Years Following Initial Vaccination in Adults Who Participated in Trial MTA29
Brief Title: Antibody Persistence and Response to Re-vaccination With Either Menactra® or Menomune® 3 Years After Initial Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA75; U1111-1115-6685 (Other: WHO)
Record Dates: First submitted 2010-11-08; First posted 2010-11-11 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Meningitis; Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningitis; Meningococcal Meningitis; Meningococcal Infections; Menactra®; Menomune®; Meningococcal vaccine
MeSH Terms: conditions — Meningitis; Meningitis, Meningococcal; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menomune® vaccine group (Experimental): Participants received Menomune® vaccine in MTA29 (NCT00874549)
  Interventions: Biological: Menomune®: A, C, Y, W 135 Meningococcal Polysaccharide
- Menactra® vaccine group (Experimental): Participants received Menactra® vaccine in trial MTA29 (NCT00874549)
  Interventions: Biological: Menactra®: Meningococcal (A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Menomune®: A, C, Y, W 135 Meningococcal Polysaccharide — 0.5 mL, Subcutaneous
  Other Names: Menomune®
  Arms: Menomune® vaccine group
Biological: Menactra®: Meningococcal (A, C, Y and W 135) Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® vaccine group

SUMMARY:
The purpose of this trial is to describe antibody persistence and response to re-vaccination with either Menactra® or Menomune® vaccine approximately three years following initial vaccination in adults who participated in trial MTA29 (NCT00874549).

Objectives:

* To describe the rates of immediate reactions, solicited injection-site and systemic reactions, all unsolicited adverse events, and serious adverse events following vaccination.
* To evaluate persistence of serum bactericidal antibodies in subjects who received Menactra® or Menomune® vaccine approximately three years ago.
* To evaluate the immune response to serogroups A, C, Y, and W-135 in subjects re-vaccinated with either Menactra® or Menomune® vaccine.

DETAILED DESCRIPTION:
Participants who were randomized and received either Menactra® or Menomune® vaccine in trial MTA29 will receive 1 dose of either Menactra® or Menomune®, respectively on Day 0 and will be followed-up for 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 56 years or older on the day of inclusion.
* Received the appropriate Menactra or Menomune vaccine as assigned by randomization in Trial MTA29.
* Ambulatory and healthy, as determined by medical history.
* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman of childbearing potential, use of an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination.

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Known pregnancy, or a positive pregnancy test.
* Currently breastfeeding a child.
* History of documented invasive meningococcal disease.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial vaccination.
* Planned participation in another clinical trial during the present trial period.
* Receipt of any meningococcal vaccine since participation in trial MTA29.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination, except for influenza vaccination, which may be received at least two weeks before trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the trial vaccination.
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Laboratory-confirmed seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B, or Hepatitis C.
* Previous personal history of Guillain-Barré Syndrome (GBS).
* Known systemic hypersensitivity to any of the vaccine components, latex, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
* Laboratory-confirmed thrombocytopenia, contraindicating intramuscular (IM) vaccination.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug use that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Not available for the entire study period or unable to attend the scheduled visits or to comply with the study procedures.
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Identified as employees of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as family members (i.e., immediate, husband, wife and their children, adopted or natural) of the employees or the Investigator.

Min Age: 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (6):
- United States (6):
  - Scottsdale, Arizona
  - Bardstown, Kentucky
  - Albuquerque, New Mexico
  - West Jordan, Utah
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 08 November 2010 to 16 December 2010 at 6 US clinical centers.
Pre-assignment Details: A total of 139 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Menomune® Vaccine Group: All participants had received Menomune® vaccine in Study MTA29 and received a single dose of Menomune® on Day 0 in the present trial.
- Menactra® Vaccine Group: All participants had received Menactra® vaccine in Study MTA29 and received a single dose of Menactra® on Day 0 in the present trial.
Period: Overall Study
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Started | 36 (For safety analysis number includes 1 participant randomized to Menactra who received Menomune.) | 103
Completed | 34 | 102
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group | Total
Number analyzed (Participants) | 36 | 103 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 28 | 36
  >=65 years | 28 | 75 | 103
Age Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (7.2) | 71.1 (6.8) | 71.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 57 | 77
  Male | 16 | 46 | 62
Region of Enrollment [Number; unit: Participants]
  United States | 36 | 103 | 139

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site or Systemic Reactions Following Vaccination With Either Menomune or Menactra Vaccine
Description: Solicited Injection Site Reactions: Pain, Erythema, Swelling. Solicited Systemic Reactions: Fever (Temperature), Headache, Malaise, Myalgia.
  Grade 3 reactions were defined as: Pain, headache, malaise, and myalgia - significant, prevents daily activity; Erythema and swelling - > 100 mm; Fever, temperature of ≥ 39.0ºC or ≥ 102.1ºF.
Time Frame: Day 0 to Day 7 post-vaccination
Population: Solicited reactions were assessed in all subjects who received at a dose of study vaccine, according to the vaccine actually received (Safety Analysis Population).
Measure: Number; unit: Participants
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 34 | 103
Participants
  Any Pain | 8 | 33 [0 to 0]
  Grade 3 Pain | 0 | 1 [0 to 0]
  Any Erythema | 9 | 0 [0 to 0]
  Grade 3 Erythema | 0 | 0 [0 to 0]
  Any Swelling | 1 | 2 [0 to 0]
  Grade 3 Swelling | 0 | 0 [0 to 0]
  Any Fever | 0 | 0 [0 to 0]
  Grade 3 Fever | 0 | 0 [0 to 0]
  Any Headache | 8 | 16 [0 to 0]
  Grade 3 Headache | 1 | 1 [0 to 0]
  Any Malaise | 3 | 8 [0 to 0]
  Grade 3 Malaise | 0 | 0 [0 to 0]
  Any Myalgia | 6 | 22 [0 to 0]
  Grade 3 Myalgia | 1 | 1 [0 to 0]

2. Other Pre Specified Outcome: Geometric Mean Titers of Individual Antibodies to Vaccine Antigens Following Vaccination With Either Menomune or Menactra Vaccine
Description: Geometric mean titers (GMTs) of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with human complement (SBA-HC).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: GMTs were assessed in participants who met all inclusion, but no exclusion criteria; received assigned study vaccine; and had serology samples with valid test results (Per-Protocol Population).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 32 | 99
Titers
  Serogroup A Pre-vaccination (N = 32, 99) | 7.2 [4.4 to 11.8] | 10.1 [7.6 to 13.3]
  Serogroup A Post-vaccination (N = 31, 99) | 15.6 [9.2 to 26.5] | 87.1 [62.0 to 122.3]
  Serogroup C Pre-vaccination (N = 32, 99) | 9.9 [5.5 to 18.0] | 6.6 [4.9 to 8.9]
  Serogroup C Post-vaccination (N = 32, 99) | 14.4 [7.4 to 27.8] | 93.4 [63.0 to 138.5]
  Serogroup Y Pre-vaccination (N = 32, 99) | 7.2 [4.1 to 12.6] | 6.2 [4.4 to 8.7]
  Serogroup Y Post-vaccination (N = 31, 99) | 11.4 [6.2 to 21.1] | 96.1 [62.1 to 148.5]
  Serogroup W-135 Pre-vaccination (N = 32, 99) | 4.1 [2.9 to 5.7] | 7.6 [5.6 to 10.4]
  Serogroup W-135 Post-vaccination (N = 31, 99) | 6.4 [4.4 to 9.3] | 80.1 [55.0 to 116.5]

3. Other Pre Specified Outcome: Summary of Participants Antibody Titers for Each of the Vaccine Serogroups Before and 28 Days After Vaccination With Either Menomune or Menactra Vaccine.
Description: Titers of antibodies to serogroups A, C, Y, and W-135 for each participant were measured by serum bactericidal assay with human complement (SBA-HC).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Antibody titers were assessed in participants who met all inclusion, but no exclusion criteria; received assigned study vaccine; and had serology samples with valid test results (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 32 | 99
Participants
  Serogroup A ≥ 1:4 Pre-vaccination (N = 32, 99) | 23 | 79 [0 to 0]
  Serogroup A ≥ 1:8 Pre-vaccination (N = 32, 99) | 14 | 57 [0 to 0]
  Serogroup A ≥ 1:4 Post-vaccination (N = 31, 99) | 28 | 97 [0 to 0]
  Serogroup A ≥ 1:8 Post-vaccination (N = 31, 99) | 24 | 92 [0 to 0]
  Serogroup C ≥1:4 Pre-vaccination (N = 32, 99) | 20 | 55 [0 to 0]
  Serogroup C ≥ 1:8 Pre-vaccination (N = 32, 99) | 17 | 41 [0 to 0]
  Serogroup C ≥1:4 Post-vaccination (N = 32, 99) | 24 | 95 [0 to 0]
  Serogroup C ≥ 1:8 Post-vaccination (N = 32, 99) | 18 | 90 [0 to 0]
  Serogroup Y ≥ 1:4 Pre-vaccination (N = 32, 99) | 15 | 43 [0 to 0]
  Serogroup Y ≥ 1:8 Pre-vaccination (N = 32, 99) | 14 | 34 [0 to 0]
  Serogroup Y ≥1:4 Post-vaccination (N = 31, 99) | 19 | 89 [0 to 0]
  Serogroup Y≥1:8 Post -vaccination (N = 31, 99) | 18 | 87 [0 to 0]
  Serogroup W-135 ≥1:4 Pre-vaccination (N = 32, 99) | 15 | 59 [0 to 0]
  Serogroup W-135 ≥1:8 Pre-vaccination (N = 32, 99) | 12 | 44 [0 to 0]
  Serogroup W-135 ≥1:4 Post-accination (N = 31, 99) | 25 | 95 [0 to 0]
  Serogroup W-135 ≥1:8 Post-vaccination (N = 31, 99) | 14 | 92 [0 to 0]

4. Other Pre Specified Outcome: Number of Participants Who Achieved a Four-Fold Rise in Bactericidal Antibody Titers From Baseline Following Vaccination With Either Menomune or Menactra Vaccine.
Description: Titers of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with human complement (SBA-HC).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 32 | 99
Participants
  Serogroup A (N = 31, 99) | 8 | 70 [0 to 0]
  Serogroup C (N = 32, 99) | 5 | 77 [0 to 0]
  Serogroup Y (N = 31, 99) | 4 | 75 [0 to 0]
  Serogroup W-135 (N = 31, 99) | 2 | 73 [0 to 0]

5. Other Pre Specified Outcome: Geometric Mean Titers of Individual Antibodies to Vaccine Antigens Following Vaccination With Either Menomune or Menactra Vaccine (SBA-BR)
Description: Geometric mean titers (GMTs) of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with baby rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 32 | 99
Titers
  Serogroup A Pre-vaccination (N = 32, 99) | 22.1 [9.5 to 51.6] | 20.2 [12.8 to 31.7]
  Serogroup A Post -vccination (N = 31, 98) | 119.7 [45.9 to 312.3] | 396.9 [266.8 to 590.5]
  Serogroup C Pre-vaccination (N = 32, 99) | 39.7 [16.2 to 97.6] | 35 [22.1 to 55.6]
  Serogroup C Post-vaccination (N = 31, 98) | 109.5 [40.2 to 298.0] | 698.9 [450.4 to 1084.7]
  Serogroup Y Pre-vaccination (N = 32, 99) | 71.3 [36.1 to 140.9] | 70.6 [46.6 to 106.8]
  Serogroup Y Post-vaccination (N = 31, 99) | 200.2 [98.8 to 405.4] | 556.9 [370.6 to 836.8]
  Serogroup W-135 Pre-vaccination (N = 32, 99) | 74.5 [37.5 to 147.9] | 79 [52.4 to 118.9]
  Serogroup W-135 Post-vaccination (N = 31, 98) | 214.1 [101.6 to 451.2] | 534.2 [351.7 to 811.4]

6. Other Pre Specified Outcome: Number of Participants With Antibody Titers at ≥ 1:8 for Each of the Vaccine Serogroups Before and After Vaccination With Either Menomune or Menactra Vaccine
Description: Titers of antibodies to vaccine serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with baby rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Antibody titers were assessed in participants who met all inclusion, but no exclusion criteria; received assigned study vaccine and serology samples with valid test results (Per-Protocol Population).
Measure: Number; unit: Participants
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 32 | 99
Participants
  Serogroup A Pre-vaccination (N = 32, 99) | 12 | 35 [0 to 0]
  Serogroup A Post-vaccination (N = 31, 98) | 21 | 87 [0 to 0]
  Serogroup C Pre-vaccination (N = 32, 99) | 17 | 53 [0 to 0]
  Serogroup C Post-vaccination (N = 31, 98) | 20 | 91 [0 to 0]
  Serogroup Y Pre-vaccination (N = 32, 99) | 26 | 75 [0 to 0]
  Serogroup Y Post-vaccination (N = 31, 99) | 29 | 94 [0 to 0]
  Serogroup W-135 Pre-vaccination (N = 32, 99) | 25 | 75 [0 to 0]
  Serogroup W-135 Post-vaccination (N = 31, 98) | 27 | 91 [0 to 0]

7. Other Pre Specified Outcome: Number of Participants Who Achieved a Four-Fold Rise in Bactericidal Antibody Titers From Baseline After Vaccination With Either Menomune or Menactra Vaccine
Description: Titers of antibodies to serogroups A, C, Y, and W-135 were measured by serum bactericidal assay with baby rabbit complement (SBA-BR).
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Number analyzed (Participants) | 31 | 99
Participants
  Serogroup A (N = 31, 98) | 12 | 69 [0 to 0]
  Serogroup C (N = 31, 98) | 10 | 78 [0 to 0]
  Serogroup Y (N = 31, 99) | 17 | 60 [0 to 0]
  Serogroup W-135 (N = 31, 98) | 13 | 67 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from vaccination on Day 0 through Day 28 post-vaccination.
Arm/Group | Menomune® Vaccine Group | Menactra® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/103
Other Adverse Events (participants affected / at risk) | 9/36 | 33/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Menomune® Vaccine Group (N=36) | Menactra® Vaccine Group (N=103)
Injection Site Pain (General disorders) | 8/34 (8) | 33 (33)
Injection Site Erythema (General disorders) | 9/34 (9) | 0 (0)
Malaise (General disorders) | 3/34 (3) | 8 (8)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6/34 (6) | 22 (22)
Headache (Nervous system disorders) | 8/34 (8) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.